CLINICAL TRIAL: NCT03842306
Title: End-tidal Oxygen Can Reliably Predict the Arterial Partial Pressure of Oxygen Among Emergency Department Patients Undergoing Rapid Sequence Intubation
Brief Title: End-tidal Oxygen Can Reliably Predict the Arterial Partial Pressure of Oxygen Among Emergency Department Patients
Status: Completed | Type: Observational
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: 17-031
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Intubation Complication
Keywords: End tidal oxygen; Preoxygenation; Arterial oxygen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: Patients undergoing rapid sequence intubation in the emergency department for which end tidal oxygen was monitored.

SUMMARY:
Recent studies have shown that end tidal oxygen (ETO2) monitoring can be useful to determine the adequacy of preoxygenation. No study has assessed the correlation between ETO2 values obtained during preoxygenation to predict the PaO2 in patients undergoing RSI in the ED. Our objective was to determine whether a novel equation using the ETO2 at the end of preoxygenation could reliably estimate the partial pressure of arterial oxygen (PaO2) in critically-ill ED patients undergoing RSI.

DETAILED DESCRIPTION:
Rapid Sequence Intubation (RSI) is the preferred and most commonly-used method of definitive airway management among critically ill emergency department (ED) patients requiring intubation. Adequate preoxygenation is intended to prolong the safe apnoeic period. Optimal preoxygenation for ED patient undergoing RSI is best described as a two-part process of denitrogenation of the functional residual capacity (FRC) and the formation of an oxygen reservoir within the alveoli. End-tidal O2 (EtO2) has been shown to be a reliable surrogate marker for denitrogenation. Most of the literature supporting EtO2 as an adequate maker of adequate preoxygenation has been conducted in the operating room setting. This population varies significantly from the population requiring endotracheal intubation in the ED. Our study aim was to show that the use of a gas analyzer measuring the fraction of inspired oxygen (FiO2) and EtO2 during the preoxygenation phase of ED RSI can reliably predict the minimal PaO2 at the end of the ED preoxygenation period.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing rapid sequence intubation.

Exclusion Criteria:

* Patients presenting to the emergency department in cardiac or traumatic arrest
* Patients who received bi-level positive airway pressure (BiPAP) as the primary delivery of preoxygenation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Emergency department patients with a need for endotracheal intubation.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Correlation of ETO2 to arterial oxygen | within 2 minutes of rapid sequence intubation
  To determine whether a novel equation using the EtO2 measured by a gas analyzer at the time of induction during the preoxygenation phase of ED RSI could reliably estimate the minimal PaO2 in patients undergoing RSI.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Caputo, MD, Principal Investigator — NYC H+H/Lincoln
Locations (1):
- NYC H+H/Lincoln, The Bronx, New York, United States

REFERENCES:
- [Background] Brown CA 3rd, Bair AE, Pallin DJ, Walls RM; NEAR III Investigators. Techniques, success, and adverse events of emergency department adult intubations. Ann Emerg Med. 2015 Apr;65(4):363-370.e1. doi: 10.1016/j.annemergmed.2014.10.036. Epub 2014 Dec 20. PMID 25533140
- [Background] Sakles JC. Maintenance of Oxygenation During Rapid Sequence Intubation in the Emergency Department. Acad Emerg Med. 2017 Nov;24(11):1395-1404. doi: 10.1111/acem.13271. Epub 2017 Oct 13. No abstract available. PMID 28791775
- [Background] Benumof JL, Dagg R, Benumof R. Critical hemoglobin desaturation will occur before return to an unparalyzed state following 1 mg/kg intravenous succinylcholine. Anesthesiology. 1997 Oct;87(4):979-82. doi: 10.1097/00000542-199710000-00034. No abstract available. PMID 9357902
- [Background] Weingart SD, Levitan RM. Preoxygenation and prevention of desaturation during emergency airway management. Ann Emerg Med. 2012 Mar;59(3):165-75.e1. doi: 10.1016/j.annemergmed.2011.10.002. Epub 2011 Nov 3. PMID 22050948
- [Background] Benumof JL. Preoxygenation: best method for both efficacy and efficiency. Anesthesiology. 1999 Sep;91(3):603-5. doi: 10.1097/00000542-199909000-00006. No abstract available. PMID 10485765
- [Background] Campbell IT, Beatty PC. Monitoring preoxygenation. Br J Anaesth. 1994 Jan;72(1):3-4. doi: 10.1093/bja/72.1.3. No abstract available. PMID 8110546
- [Background] Bhatia PK, Bhandari SC, Tulsiani KL, Kumar Y. End-tidal oxygraphy and safe duration of apnoea in young adults and elderly patients. Anaesthesia. 1997 Feb;52(2):175-8. doi: 10.1111/j.1365-2044.1997.14-az016.x. PMID 9059106
- [Background] Farmery AD, Roe PG. A model to describe the rate of oxyhaemoglobin desaturation during apnoea. Br J Anaesth. 1996 Feb;76(2):284-91. doi: 10.1093/bja/76.2.284. PMID 8777112
- [Background] Groombridge C, Chin CW, Hanrahan B, Holdgate A. Assessment of Common Preoxygenation Strategies Outside of the Operating Room Environment. Acad Emerg Med. 2016 Mar;23(3):342-6. doi: 10.1111/acem.12889. Epub 2016 Feb 17. PMID 26728311
- [Background] Bodily JB, Webb HR, Weiss SJ, Braude DA. Incidence and Duration of Continuously Measured Oxygen Desaturation During Emergency Department Intubation. Ann Emerg Med. 2016 Mar;67(3):389-95. doi: 10.1016/j.annemergmed.2015.06.006. Epub 2015 Jul 9. PMID 26164643
- [Background] Mort TC. Preoxygenation in critically ill patients requiring emergency tracheal intubation. Crit Care Med. 2005 Nov;33(11):2672-5. doi: 10.1097/01.ccm.0000187131.67594.9e. PMID 16276196
- [Background] Mort TC. The incidence and risk factors for cardiac arrest during emergency tracheal intubation: a justification for incorporating the ASA Guidelines in the remote location. J Clin Anesth. 2004 Nov;16(7):508-16. doi: 10.1016/j.jclinane.2004.01.007. PMID 15590254
- [Background] Mosier JM, Hypes CD, Sakles JC. Understanding preoxygenation and apneic oxygenation during intubation in the critically ill. Intensive Care Med. 2017 Feb;43(2):226-228. doi: 10.1007/s00134-016-4426-0. Epub 2016 Jun 24. No abstract available. PMID 27342820